CLINICAL TRIAL: NCT01168115
Title: Near-Infrared Spectroscopy for Blood Glucose Measurements
Status: Completed | Type: Observational
Sponsor: InLight Solutions (Industry)
Collaborators: Luminous Medical (Industry)
Responsible Party: Ries Robinson, InLight
Other Study IDs: ILS-07-386
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2008-01

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this study is to evaluate the performance of a near-infrared transmission measurement in blood samples collected from healthy volunteers. We propose that NIR spectroscopic blood glucose measurements in healthy patients are as accurate as handheld glucometers and a Yellow Springs Instrument (YSI). We will also evaluate in vitro blood samples spiked with pharmacological interferents to test if the spectroscopic glucose measurement is affected by common medications.

DETAILED DESCRIPTION:
Luminous Medical is developing an automated glucose measurement system that addresses the rapidly growing clinical demand for tight glycemic control in the intensive care unit (ICU), operating room (OR), and intermediate care units. The system automatically measures glucose and other analytes by spectroscopically analyzing blood as it passes through a disposable Sensor Set. Our unique optical measurement does not chemically interact with blood, is insensitive to sensor fouling, and, unlike a biosensor, does not require frequent recalibration.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 and 65
* Healthy
* Not currently pregnant
* Hematocrit >38%

Exclusion Criteria:

* Pregnancy (Self Reported)
* Females that have given birth 6 weeks prior (self reported)
* Anemia (hematocrit <38%) Hematocrit is checked via a capillary fingerstick and a blood hematocrit reader.
* Under the age of 18 or over the age of 65.
* Diagnosed with Type I or II Diabetes (Self-Reported).
* Donated blood (>25 mls) in the last 8 weeks
* Heart rate >100 beats per minute
* Weigh less than 110 lbs.
* Currently taking anticoagulants (ex: coumadin)
* Abnormal blood pressure (diastolic >90)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males and females between the ages of 18 and 65
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rohrscheib, M.D., Principal Investigator — UNMHSC
Locations (1):
- InLight Solutions, Albuquerque, New Mexico, United States

REFERENCES:
- See also: Related Info — http://www.inlightsolutions.com
- See also: Related Info — http://www.luminousmedical.com